CLINICAL TRIAL: NCT06136546
Title: The Role of Inflammation in Cognitive Dysfunction in Acute Depression as Determined by Experimental Inhibition of Tumor Necrosis Factor-alpha Signaling in a Randomized Controlled Trial.
Brief Title: Cognitive Dysfunction and Inflammation in Depression: Experimental Inhibition Via Infliximab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Naoise Mac Giollabhui, PhD, Member of the Faculty, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023p002988
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Depressive Disorder, Major; Inflammation
Keywords: Depression; Major Depressive Disorder; Infliximab; Cognitive Dysfunction
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation; Depression; Cognitive Dysfunction | interventions — Infliximab

STUDY DESIGN:
Intervention Model Description: A permuted block design (n=4) on a 1:1 allocation will be used to assign participants to each intervention group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All treatment teams, outcome assessors, and data analysts will be blind to randomization assignment until the primary study results have been analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Infliximab (Experimental): Participants in this arm will receive 5 mg/kg of infliximab via an in-dwelling catheter.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Participants in this arm will receive saline as placebo via an in-dwelling catheter.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Infliximab — Intravenous infusion of infliximab
  Arms: Infliximab
Other: Placebo — Intravenous infusion of saline solution (matching in color and consistency in infliximab)
  Arms: Placebo

SUMMARY:
This study is a mechanistic randomized controlled trial that investigates whether inhibition of tumor necrosis factor signaling via intravenous infusion of infliximab improves psychomotor speed and executive functioning in depressed individuals who exhibit an inflammatory phenotype.

DETAILED DESCRIPTION:
In this mechanistic RCT, depressed adults who exhibit a pro-inflammatory phenotype (C reactive protein ≥3mg/L) will be randomized on a 1:1 allocation to receive a TNF inhibitor (infliximab) or placebo. Over a two-week follow-up, participants will remotely complete brief, daily assessments of depressive symptoms and psychomotor speed/executive functioning using a mobile-based platform (TestMyBrain) in addition to in-person clinician-rated assessment of depressive symptom severity (Hamilton Depression Rating Scale), anhedonia (Dimensional Anhedonia Rating Scale), and more comprehensive computerized batteries assessing cognitive function (TestMyBrain). Blood will be drawn at baseline and week 1 to assess immune biomarkers (C reactive protein, tumor necrosis factor- alpha and its soluble receptors). Specifically, the study will determine whether randomization to infliximab is associated with improvement in psychomotor speed and executive function.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 25-50 years
2. Able to read and understand English and willing to provide informed consent/comply with the study protocol
3. Willingness to complete intravenous infusion and have blood drawn
4. Exhibit circulating blood level of C reactive protein ≥ 3mg/L
5. Diagnosed with Major Depressive Disorder
6. Moderate depressive symptom severity, as indicated by score ≥15 on the Hamilton Depression Rating Scale
7. Antidepressant treatment free for at least 4 weeks prior to study entry or be on a fixed treatment regimen for at least 4 weeks; willingness to continue treatment status (i.e., change/begin new treatment) until study termination
8. Willingness not to begin/change therapies until study termination (maximum of three weeks following screening)
9. Be of non-childbearing potential per the following specific criteria:

   a. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or b. Childbearing potential and meets the following criteria: i. A negative serum pregnancy test within thirty days of infusion (may be repeated closer to infusion date at the discretion of the PI or study staff) and abstinent after the negative serum pregnancy test and prior to infusion; or ii. Using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent; iii. Continuously use one of the following methods of birth control over the last six months: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence.

Exclusion Criteria:

1. Medical conditions that could confound interpretation or increase participant risk, as indicated via medical history or laboratory testing; exclusionary medical conditions will include:

   i. acute injury/infection within one week of study initiation or infection within one month of study initiation that required antibiotic/antiviral treatment ii. chronic infection (e.g., hepatitis B or C or HIV) or history of Covid 19 infection within the past 6 months or with persisting symptoms.

   iii. latent infection (e.g., tuberculosis, fungal infections), or history of recurrent infections, iv. uncontrolled cardiovascular, endocrine, hematologic, hepatic, renal or neurologic disease (as determined by medical history, physical exam and laboratory testing) v. cancer history vi. autoimmune conditions; neurologic conditions (controlled) that are known to substantially impact cognitive function (e.g., stroke).

   Of note, stable medical conditions such as diabetes and cardiovascular disease, will be allowed in the study as they can contribute to endogenous inflammation.
2. Active antipsychotic and anticonvulsant medication use (that interact with infliximab)
3. Prior use of a TNF antagonist or use of systemic corticosteroids or anti-proliferative agents within one year of study entry
4. History of liver abnormalities
5. Major cognitive impairment as determined by study investigators
6. Active restrictive eating disorder or obsessive compulsive disorder deemed by study investigators to be primary cause of depressive disorder
7. History of a psychotic disorder or Bipolar disorder type I/II
8. Current substance use disorder (i.e., present in last six months), of greater than mild severity
9. Suicidal ideation based on a score ≥3 on the Columbia-Suicide Severity Rating Scale
10. Electroconvulsive therapy (ECT)/deep brain stimulation (DBS) within the last year, or report of persistent negative cognitive effects of ECT/DBS
11. Presence of a transplanted solid organ
12. Medication use affecting immune or cognitive function:

    i. Chronic use (>1 month) of a benzodiazepine more than the equivalent of 2 mg of lorazepam ii. Use of anti-inflammatory agents during the study: non-steroidal anti-inflammatory agents (NSAIDs) (excluding 81mg of aspirin), glucocorticoid containing medicines or statins, or cyclooxygenase-2 (COX-2) inhibitors
13. Considered by the study investigators to be inappropriate for the study due to safety concerns or to be unlikely to complete the protocol
14. History of allergic response to murine products

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Speed (TestMyBrain: Simple Reaction Time) | Repeated measures over two weeks
  Faster within-person psychomotor speed (i.e. median response time)
Executive Function (TestMyBrain: Choice Reaction Time) | Repeated measures over two weeks
  Better within-person executive function performance (i.e. accuracy-adjusted response speed)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (17-item; range 0-54) | Week 2
  Reduced depressive symptoms severity
Dimensional Anhedonia Rating Scale (17-item; range 0-68) | Week 2
  Reduced anhedonia
Concentrations of circulating C reactive protein | Week 1
  Reduced circulating C reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No